CLINICAL TRIAL: NCT07110220
Title: All-ceramic Restorations on Teeth and Implants: Retrospective and Prospective Study
Brief Title: All-ceramic Restorations: a Retrospective and Prospective Study
Acronym: PROCER
Status: Enrolling by invitation | Type: Observational
Sponsor: Mainjot Amélie (Other)
Responsible Party: Sponsor-Investigator, Mainjot Amélie, Professor, Centre Hospitalier Universitaire de Liege
Organization: Centre Hospitalier Universitaire de Liege (Other)
Other Study IDs: B7072024000038
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Tooth Disorder; Missing Tooth/Teeth
MeSH Terms: conditions — Tooth Diseases; Anodontia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to evaluate the survival and success rate of ceramic restorations on teeth and implants done in the department of fixed prosthodontics at the CHU of Liege for the last 25 years.

The main question it aims to answer is: Are ceramic restorations reliable and sustainable ?

Participants already treated with ceramic restoration will answer survey questions about their restoration once a year, in parallel with clinical evaluation following Hickel et al 2010 (Science Committee of the FDI World Dental Federation -FDI) to assess esthetic, functional, mechanical and biological properties of the restorations .

ELIGIBILITY:
Inclusion Criteria:

* The study population consists of patients attending the dentistry department of the University Hospital of Liège who have had ceramic restorations fitted by one of the practitioners in the fixed prosthetics department of the University Hospital of Liège over the last 25 years.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients attending the dentistry department of the University Hospital of Liège who have had ceramic restorations fitted by one of the practitioners in the fixed prosthetics department of the University Hospital of Liège over the last 25 years.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2039-06-15 (Estimated); Study Completion 2039-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation of ceramic restoration on teeth and implants | 15 years
  Clinical evaluation following FDI criteria

SECONDARY OUTCOMES:
Satisfaction evaluation of patient with ceramic restoration | 15 years
  Satisfaction questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital (CHU) of Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hickel R, Peschke A, Tyas M, Mjor I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation - clinical criteria for the evaluation of direct and indirect restorations. Update and clinical examples. J Adhes Dent. 2010 Aug;12(4):259-72. doi: 10.3290/j.jad.a19262. PMID 20847997